CLINICAL TRIAL: NCT01773395
Title: A Randomized Placebo-controlled Phase II Trial of Irradiated, Adenovirus Vector Transferred GM-CSF Secreting Autologous Leukemia Cell Vaccination (GVAX) Versus Placebo Vaccination in Patients With Advanced MDS/AML After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: GVAX vs. Placebo for MDS/AML After Allo HSCT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recommendation by the Data and Safety Monitoring Board due to efficacy concerns
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Vincent T. Ho, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-217
Record Dates: First submitted 2013-01-08; First posted 2013-01-23 (Estimated); Results first posted 2022-03-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-06

CONDITIONS: Myelodysplastic Syndrome; Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia
Keywords: Advanced
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic | interventions — Busulfan; fludarabine; Tacrolimus; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GVAX (Active Comparator): GVAX vaccine
  Participants in the GVAX vaccine arm will undergo a conditioning regimen with busulfan and fludarabine prior to allogeneic hematopoietic stem cell transplant. Immediately after allogeneic hematopoietic stem cell transplant participants will start tacrolimus and methotrexate to prevent GVHD. GVAX arm participants meeting criteria to begin vaccinations will be administered the GVAX vaccine at established study time points.
  Interventions: Biological: GVAX; Procedure: Allogeneic Hematopoietic Stem Cell Transplant; Drug: Busulfan; Drug: Fludarabine; Drug: Tacrolimus; Drug: Methotrexate
- Placebo (Placebo Comparator): Placebo vaccine
  Participants in the Placebo vaccine arm will undergo a conditioning regimen with busulfan and fludarabine prior to allogeneic hematopoietic stem cell transplant. Immediately after allogeneic hematopoietic stem cell transplant participants will start tacrolimus and methotrexate to prevent GVHD. Placebo vaccine arm participants meeting criteria to begin vaccinations will be administered the placebo vaccine at established study time points.
  Interventions: Biological: Placebo Vaccine; Procedure: Allogeneic Hematopoietic Stem Cell Transplant; Drug: Busulfan; Drug: Fludarabine; Drug: Tacrolimus; Drug: Methotrexate

INTERVENTIONS:
Biological: GVAX — GVAX or placebo vaccination will begin between 30 to 60 days following participant's transplant, provided participant meets vaccination initiation criteria. Only participants in the GVAX arm will receive GVAX vaccine.
  Arms: GVAX
Biological: Placebo Vaccine — GVAX or placebo vaccination will begin between 30 to 60 days following participant's transplant, provided participant meets vaccination initiation criteria. Only participants in the placebo arm will receive placebo vaccine.
  Arms: Placebo
Procedure: Allogeneic Hematopoietic Stem Cell Transplant — Between 1-2 days after participant finishes the chemotherapy, the participant will receive the blood stem cell or marrow from their donor. This is given as a transfusion through a central intravenous line (IV usually placed in the chest or arm).
Drug: Busulfan — In this study the condition regimen will include 2 chemotherapy drugs: busulfan (twice a day or four times a day for 5 days) and fludarabine (once daily for 4 days). Depending on participant's age, and other clinical factors, the transplant doctor will decide whether the participant will receive a higher or lower dose of busulfan.
Drug: Fludarabine — In this study the condition regimen will include 2 chemotherapy drugs: busulfan (twice a day or four times a day for 5 days) and fludarabine (once daily for 4 days). Depending on participant's age, and other clinical factors, the transplant doctor will decide whether the participant will receive a higher or lower dose of busulfan.
Drug: Tacrolimus — Just prior to and immediately following the infusion of stem cells, the participant will receive medications to help prevent graft-versus-host disease (GVHD), a common complication of transplant where the donor's immune cells attack the recipient's body. The medications the participant will receive to prevent GVHD will include:
  * Tacrolimus- This will be taken orally twice daily start 3 days before the transplant, and will continue for about 6-9 months.
  * Methotrexate- This will be given a short intravenous infusion on days 1, 3, 6, and 11 after the transplant.
Drug: Methotrexate — Just prior to and immediately following the infusion of stem cells, the participant will receive medications to help prevent graft-versus-host disease (GVHD), a common complication of transplant where the donor's immune cells attack the recipient's body. The medications the participant will receive to prevent GVHD will include:
  * Tacrolimus- This will be taken orally twice daily start 3 days before the transplant, and will continue for about 6-9 months.
  * Methotrexate- This will be given a short intravenous infusion on days 1, 3, 6, and 11 after the transplant.

SUMMARY:
This research study is a Phase II clinical trial. Phase II clinical trials test the effectiveness of an investigational intervention to learn whether the intervention, in this case, the GVAX vaccine, works in preventing MDS, CMML, or AML from relapsing after allogeneic stem cell transplantation. "Investigational" means that the vaccine is still being studied and that research doctors are trying to find out more about it-such as the side effects it may cause, and if the vaccine is effective. It also means that the FDA has not yet approved the vaccine for these types of cancer.

Participants are being asked to participate in this trial because they have advanced myelodysplastic syndrome (MDS), Chronic Myelomonocytic Leukemia (CMML), or acute myeloid leukemia (AML). Investigators have determined that participants are a candidate for an allogeneic stem cell transplant as treatment for MDS/CMML/AML. Allogeneic stem cell transplantation is a standard treatment for MDS/CMML/AML. It can be effective because the cells from the donor (also known as the graft) could form a new immune system that can fight against the MDS/CMML/AML cells in the body. This is also known as the "graft-versus-leukemia" or "GVL" effect. In patients with advanced MDS, CMML, or AML that is not in remission at the time of transplantation, relapse remains the number one cause of transplant failure. As such, this clinical trial is designed to assess whether adding a leukemia vaccine early after transplantation could stimulate donor cells to fight cancer and improve transplant outcomes.

In recent years, researchers at the Dana-Farber Cancer Institute have discovered that GVAX, a vaccine made from the patient's own cancer cells engineered to produce a protein called GM-CSF, can be effective in stimulating a powerful immune response specific to that cancer. GM-CSF is a naturally occurring hormone in the body that helps the immune system fight infections and diseases. The GVAX vaccine is made in the laboratory by using a virus (called adenovirus, which has been modified so it cannot cause illness) to insert the GM-CSF gene into tumor cells. The cells are then irradiated, which prevents them from being able to grow, before being administered to patients in a series of vaccinations.

A previous phase I clinical trial using this GVAX vaccine in patients with MDS/AML after allogeneic transplantation demonstrated that the GVAX vaccine is safe, and the survival outcomes were encouraging. The current randomized phase II study will investigate this vaccine further and gather more information to assess the activity.

Participants in this study will be "randomized" to receive either GVAX vaccination or placebo (a saline solution) vaccination. Randomization means participants are put into a group by chance. It is like flipping a coin. There is a 50% chance they will receive the GVAX vaccine and a 50% chance they will receive placebo. Neither participants nor investigators will know which participants will be receiving.

The primary goal of this trial is to assess if there will be a difference in the percentage of cancer free survivors in the vaccinated vs. placebo group at 18 months after transplant.

DETAILED DESCRIPTION:
This trial can be divided into four phases: 1) Pre-Transplant; 2) Allogeneic Transplant; 3) Vaccination; and 4) Post-Vaccination Follow-Up.

Phase 1: Pre-Transplant After signing the consent form participants will undergo some screening tests to find out if they can be in this research study. These tests include a medical history, physical examination, performance status, bone marrow aspirate and biopsy, blood tests, tuberculosis skin test, HLA antibody test, pregnancy test, urine test, ECHO, MUGA or RVG to measure heart function, chest x-ray, pulmonary function tests and dental consult. If these tests show that participants are eligible to participate in the research study, they will be enrolled on the trial and randomized to receive either the GVAX vaccine or the placebo vaccine after their transplant. After enrolling in the study participants will undergo additional research procedures including a blood draw and leukemia cell collection.

Phase 2: Allogeneic Transplant The transplant phase of the study will begin when participants are admitted to the hospital to receive the chemotherapy and stem cell transplant. In the week before participants receive the stem cells, they will be treated with chemotherapy. The combination of chemotherapy given before the donor cells are infused is called the conditioning regimen. The chemotherapy conditioning is given to suppress the immune system so that the donor blood stem cells will not be rejected after transplantation. The chemotherapy may also reduce the number of MDS/CMML/AML cancer cells in participants' body.

In this study the condition regimen will include 2 chemotherapy drugs: busulfan (twice a day or four times a day for 4 days) and fludarabine (once daily for 4 days). Depending on participants' age and other clinical factors, the transplant doctor will decide whether they receive a higher or lower dose of busulfan. Between 1-2 days after participants finish the chemotherapy, they will receive the blood stem cell or marrow from the donor. This is given as a transfusion through a central intravenous line (IV usually placed in the chest or arm).

Just prior to and immediately following the infusion of stem cells, participants receive medications to help prevent graft-versus-host disease (GVHD), a common complication of transplant where the donor's immune cells attack the body. The medications participants receive to prevent GVHD will include Tacrolimus and Methotrexate.

Participants will be closely monitored as per standard transplant care after their stem cell transplant. If participants received the higher dose chemotherapy conditioning, they will stay in the hospital for an average of about 3-4 weeks. If they received the lower dose conditioning transplant, their hospital admission for transplant may be shorter depending on clinical condition.

After participants' stem cell infusion, they may receive daily injections of a medication called rhGM-CSF, or Leukine, to help their white blood cells to recover faster. participants may receive this medication for up to 2 weeks. They will also be given antiviral and antibiotic medications to prevent infections as per standard practice after transplantation.

Between 20 to 30 days after stem cell infusion participants will have a physical examination, routine blood work and a blood draw for future immune tests.

Between 30 to 60 days after transplant participants will return to clinic for a visit that will include a physical examination, routine blood work, a blood draw for future immune tests and a bone marrow biopsy and aspirate to assess their MDS/CMML/AML.

Phase 3: Vaccination Participants may begin receiving the GVAX or placebo vaccination between 30 to 60 days following their transplant, provided their blood counts have recovered, and do not have any severe side effects from the transplant. If by day 61, participants' blood counts have not recovered sufficiently, or if they have developed side effects or GVHD from the transplant, and do not meet the conditions necessary to start the vaccination portion of this trial, then they will not receive any vaccinations and will be removed from the study. Participants will continue to receive standard post transplant care.

If participants are able to begin the vaccinations between day 30-60 after their transplant, the GVAX or placebo vaccine will be administered as an injection under and into the skin on the forearms or thighs, 6 times over a period of 9 weeks. The first 3 vaccinations will be administered once a week for 3 consecutive weeks and the last 3 vaccines will be given once every other week over 6 weeks. All vaccinations will be given either as an inpatient or outpatient in the clinic. On the days participants receive vaccination, they may have to wait several hours in the clinic while the laboratory makes final preparations on the vaccine/placebo.

During this 9 week period of vaccination, participants will continue to be followed by their doctor at least on a weekly basis to monitor for any transplant or possible vaccine side effects. Two to three days after the first and fifth vaccinations, investigators would encourage (but do not require) participants to return to the clinic to have a skin biopsy of the GVAX/Placebo vaccination site, especially if there is redness or swelling in the area. This will allow researchers to assess whether the new immune system is reacting to the injected leukemia cells under the microscope.

During the course of the study, investigators will also be drawing participants' blood on a regular basis to evaluate immune cells and the effect that the vaccinations may have on their new immune system.

If participants tolerate the vaccinations well, and do not have GVHD or any severe side effects from the transplant or the vaccinations, they will complete a total of 6 vaccines. However, vaccination may be terminated earlier if they develop any side effects (from transplant or vaccination) that do not resolve/improve after 2 weeks, if they develop GVHD that requires steroid treatment, or if their MDS/CMML/AML relapses and need to receive more treatment.

Phase 4: Post Vaccination Follow-Up About 1 month after the last vaccination, participants will have a physical examination, blood work, immune bloods and bone marrow biopsy and aspirate to assess the status of Their disease.

Participants will be followed at an appointment 6, 9, 12 and 18 months following their transplant with physical examinations, blood work and immune bloods. At the 12 and 18 month visit they will have a bone marrow biopsy and aspirate to assess the status of their AMLCMML//MDS.

ELIGIBILITY:
Inclusion Criteria:

* AML, CMML-with excess blasts, MDS-RAEB not in remission prior to leukemia cell harvest
* HLA 8/8 or 7/8 matched related or unrelated donor available
* ECOG performance status of 0-2
* Suitable candidate for myeloablative or reduced intensity conditioning allogeneic HSCT using PBSC or marrow as stem cell resource
* Normal organ function

Exclusion Criteria:

* Pregnant or breastfeeding
* Leukemia with active CNS involvement
* Positive HIV or HTLV-1 serology
* History of allergic reactions to compounds of similar chemical or biologic composition to GM-CSF
* Uncontrolled intercurrent illness
* History of different malignancy except if disease free for at least two years or cervical cancer in situ, basal or squamous cell carcinoma of the skin diagnosed and treated within the past two years
* Prior allogeneic transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2013-01-08 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2021-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Ho, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- [Derived] Ho VT, Kim HT, Brock J, Galinsky I, Daley H, Reynolds C, Weber A, Pozdnyakova O, Severgnini M, Nikiforow S, Cutler C, Koreth J, Alyea EP, Antin JH, Gooptu M, Romee R, Shapiro R, Chen YB, Rosenblatt J, Avigan D, Hodi FS, Dranoff G, Wu CJ, Ritz J, Soiffer RJ. GM-CSF secreting leukemia cell vaccination for MDS/AML after allogeneic HSCT: a randomized, double-blinded, phase 2 trial. Blood Adv. 2022 Apr 12;6(7):2183-2194. doi: 10.1182/bloodadvances.2021006255. PMID 34807983

RESULTS

PARTICIPANT FLOW:
Groups:
- GVAX: GVAX vaccine
  Participants in the GVAX vaccine arm will undergo a conditioning regimen with busulfan and fludarabine prior to allogeneic hematopoietic stem cell transplant. Immediately after allogeneic hematopoietic stem cell transplant participants will start tacrolimus and methotrexate to prevent GVHD.
  Conditioning regimen: In this study the condition regimen will include 2 chemotherapy drugs: busulfan (twice a day or four times a day for 4 days) and fludarabine (once daily for 4 days). Depending on participant's age, and other clinical factors, the transplant doctor will decide whether the participant will receive a higher or lower dose of busulfan.
  Allogeneic Hematopoietic Stem Cell Transplant: Between 1-2 days after participant finishes the chemotherapy, the participant will receive the blood stem cell or marrow from their donor.
  GVHD Prevention:
  * Tacrolimus- This will be taken orally twice daily start 3 days before the transplant, and will continue for about 6-9 months.
  * Methotrexate- This will be given a short intravenous infusion on days 1, 3, 6, and 11 after the transplant.
  GVAX: GVAX vaccination will begin between 30 to 45 days following participant's transplant, provided participant meets vaccination initiation criteria.
- Placebo: Placebo vaccine
  Participants in the placebo vaccine arm will undergo a conditioning regimen with busulfan and fludarabine prior to allogeneic hematopoietic stem cell transplant. Immediately after allogeneic hematopoietic stem cell transplant participants will start tacrolimus and methotrexate to prevent GVHD.
  Conditioning regimen: In this study the condition regimen will include 2 chemotherapy drugs: busulfan (twice a day or four times a day for 4 days) and fludarabine (once daily for 4 days). Depending on participant's age, and other clinical factors, the transplant doctor will decide whether the participant will receive a higher or lower dose of busulfan.
  Allogeneic Hematopoietic Stem Cell Transplant: Between 1-2 days after participant finishes the chemotherapy, the participant will receive the blood stem cell or marrow from their donor.
  GVHD Prevention:
  * Tacrolimus- This will be taken orally twice daily start 3 days before the transplant, and will continue for about 6-9 months.
  * Methotrexate- This will be given a short intravenous infusion on days 1, 3, 6, and 11 after the transplant.
  Placebo: Placebo vaccination will begin between 30 to 45 days following participant's transplant, provided participant meets vaccination initiation criteria.
Period: Overall Study
Arm/Group | GVAX | Placebo
Started | 64 | 59
Completed | 30 | 27
Not Completed | 34 | 32

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population only includes participants who received at least 1 GVAX or placebo vaccine
Groups:
- Placebo: Placebo
  Participants in the Placebo vaccine arm will undergo a conditioning regimen with busulfan and fludarabine prior to allogeneic hematopoietic stem cell transplant. Immediately after allogeneic hematopoietic stem cell transplant participants will start tacrolimus and methotrexate to prevent GVHD.
  Conditioning regimen: In this study the condition regimen will include 2 chemotherapy drugs: busulfan (twice a day or four times a day for 4 days) and fludarabine (once daily for 4 days). Depending on participant's age, and other clinical factors, the transplant doctor will decide whether the participant will receive a higher or lower dose of busulfan.
  Allogeneic Hematopoietic Stem Cell Transplant: Between 1-2 days after participant finishes the chemotherapy, the participant will receive the blood stem cell or marrow from their donor.
  GVHD Prevention:
  * Tacrolimus- This will be taken orally twice daily start 3 days before the transplant, and will continue for about 6-9 months.
  * Methotrexate- This will be given a short intravenous infusion on days 1, 3, 6, and 11 after the transplant.
  Placebo: Placebo vaccination will begin between 30 to 45 days following participant's transplant, provided participant meets vaccination initiation criteria.
- Total: Total of all reporting groups
Arm/Group | GVAX | Placebo | Total
Number analyzed (Participants) | 30 | 27 | 57
Age, Continuous [Mean (Full Range); unit: years] | 64 [27 to 75] | 63 [35 to 74] | 63 [27 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 19 | 15 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 29 | 24 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 30 | 27 | 57
Donor Age [Median (Full Range); unit: years] | 28 [19 to 67] | 30 [19 to 68] | 28 [19 to 68]
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Population: ECOG Score at baseline was not available for one participant
  Participants
    number analyzed (Participants) | 29 | 27 | 56
    ECOG 0-Fully active; no performance restrictions. | 4 | 7 | 11
    ECOG 1-Strenuous physical activity restricted; fully ambulatory and able to carry out light work. | 18 | 15 | 33
    ECOG 2-Capable of all self-care but unable to carry out any work activity Up and about >50% of time | 7 | 5 | 12
Donor Sex [Number; unit: participants]
  Female Donor | 6 | 11 | 17
  Male Donor | 24 | 16 | 40
Male Recipient With female Donor [Number; unit: participants] | 2 | 4 | 6
Disease Transplanted [Count of Participants; unit: Participants]
  Acute Myeloid Leukemia | 11 | 10 | 21
  Myelodysplastic Syndrome | 19 | 17 | 36
Acute Myeloid Leukemia Disease Status At Transplantation [Count of Participants; unit: Participants] — Population: Only patients with AML analyzed.
  Participants
    number analyzed (Participants) | 11 | 10 | 21
    2nd Complete Remission-Leukemia returned after a remission and there are now no signs of disease | 0 | 1 | 1
    Induction Failure-Leukemia has not gone away and not responded to 2 cycles of chemotherapy | 8 | 6 | 14
    Relapsed- Leukemia has returned after a period of remission | 2 | 3 | 5
    Untreated- Leukemia has never been treated | 1 | 0 | 1
AML European Leukemia Net (ELN) Risk Stratification [Count of Participants; unit: Participants] — System used to provide prognostic information in AML based on identified genetic abnormalities. Scale is from favorable to intermediate to adverse. Population: Only patients with AML analyzed
  Participants
    number analyzed (Participants) | 11 | 10 | 21
    Favorable (Best Risk) | 0 | 0 | 0
    Intermediate (Middle Risk) | 5 | 4 | 9
    Adverse (Worst Risk) | 6 | 6 | 12
Myelodysplastic Syndrome Type at Transplant [Count of Participants; unit: Participants] — Population: Only patients with MDS analyzed
  Participants
    number analyzed (Participants) | 19 | 17 | 36
    Treatment Related MDS- MDS arising from cytotoxic therapy given for a prior condition | 3 | 4 | 7
    Non-Treatment Related MDS- Disease which has arisen with no apparent cause | 16 | 13 | 29
MDS Revised International Prognostic Scoring System Risk at Transplant [Count of Participants; unit: Participants] — System used to assess the prognosis of patients with myelodysplastic syndromes. With scale of Very good to Very Poor. Population: Only patients with MDS analyzed
  Participants
    number analyzed (Participants) | 19 | 17 | 36
    Good | 10 | 8 | 18
    Intermediate | 3 | 3 | 6
    Poor | 4 | 2 | 6
    Very Poor | 2 | 4 | 6
MDS TP53 Mutated [Count of Participants; unit: Participants] — Tumor protein 53 TP53 defects influence adversely the MDS clinical outcome and the treatment response rate. Subjects were evaluated for mutations in this gene to help determine prognosis Population: Only patients with MDS analyzed
  Participants
    number analyzed (Participants) | 19 | 17 | 36
    No | 14 | 10 | 24
    Yes | 2 | 5 | 7
    Not Done | 3 | 2 | 5
Cytoreductive therapy before HSCT [Count of Participants; unit: Participants]
  No | 5 | 5 | 10
  Yes | 25 | 22 | 47
Marrow Blasts at enrollment [Median (Full Range); unit: Percent of participants] | 13 [4 to 60] | 11 [4 to 58] | 12 [4 to 60]
Donor Type [Count of Participants; unit: Participants]
  Matched Unrelated | 24 | 18 | 42
  Matched Sibling | 6 | 9 | 15
Cytomegalovirus (CMV) Serology Status [Count of Participants; unit: Participants] — Cytomegalovirus infection is a risk in this population. Prior exposure of the stem cell donor and recipient is important in determining prognosis
  Participants
    Recipient +/ Donor + | 4 | 6 | 10
    Recipient +/ Donor - | 9 | 6 | 15
    Recipient -/ Donor + | 4 | 5 | 9
    Recipient -/ Donor - | 13 | 10 | 23
Conditioning Regimen [Count of Participants; unit: Participants]
  Myeloablative Conditioning Busulfan 4 days/Fludarabine | 15 | 15 | 30
  Reduced Intensity Conditioning Busulfan 2 days/Fludarabine | 15 | 12 | 27
Graft Source [Count of Participants; unit: Participants]
  Bone Marrow | 2 | 2 | 4
  Peripheral Blood | 28 | 25 | 53

OUTCOME MEASURES:

1. Primary Outcome: 18-Month Progression Free Survival
Description: Progression-Free Survival (PFS) at 18 months after randomization. Progression-free survival is defined as time from randomization to progression of disease or death whichever occurs first. Patients with relapse/progressive disease who re-enter remission after vaccination or upon withdrawal of immune suppression alone will not be considered as having disease progression. The primary analysis will be performed using the modified intention-to-treat (ITT) principle, i.e., all transplanted and eligible patients who receive at least one vaccination will be included in the analysis according to the treatment arm they are randomized to. Patients who have not progressed and are alive are censored at the date the patient is known to be progression-free.
  Progression is defined by either morphological evidence of acute leukemia or MDS consistent with pre-transplant features
  is defined by either morphological evidence of acute leukemia or MDS consistent with pre-transplant features
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | GVAX | Placebo
Number analyzed (Participants) | 30 | 27
Percentage | 53 [34 to 69] | 55 [35 to 72]

2. Secondary Outcome: Percentage of Participants Experiencing Grade 3 or Higher Non-Hematologic or Grade 4 or Higher Hematologic Adverse Events
Description: Percentage of participants experiencing grade 3 or higher non-hematologic or grade or higher hematologic adverse events evaluated by CTCAE v5.0.
Time Frame: 18 Months
Measure: Number; unit: Percentage of participants
Arm/Group | GVAX | Placebo
Number analyzed (Participants) | 30 | 27
Percentage of participants | 3.33 | 0

3. Secondary Outcome: Percentage of Participants Experiencing Acute and Chronic Graft-Versus-Host Disease
Description: Percentage of participants with acute and chronic graft-versus-host disease (GVHD). The time frame for the acute incidence is 1 year and for chronic is 3 years.Grading of aGVHD was derived by consensus grading (Przepiorka 1995). The aGVHD algorithm calculates the grade based on the organ (skin, GI and liver) stage and etiology/biopsy reported. Skin staging: Stage 1. <25% rash; 2. 25-50%; 3. >50%; 4. generalized erythroderma with bullae. GI staging: Stage 1. Diarrhea>500ml/d or persistent nausea; 2. >1000ml/d; 3. >1500ml/d; 4. Large volume diarrhea and severe abdominal pain +- ileus. Liver staging: Stage 1. bilirubin 2-3mg/dl; 2. bili 3-6 mg/dl; 3. bili 6-15 mg/dl; 4. bili>15mg/dl. Grade 4 is the worst outcome.
  Chronic GVHD is classified using the NIH Consensus Criteria. 8 organs will be scored on a 0-3 scale to reflect degree of cGVHD involvement 0 being none, 1 mild, 2 moderate 3 severe. Liver and pulmonary function test results will also be recorded. Severe is the worst outcome
Time Frame: 1 and 3 years
Measure: Number; unit: Percentage of participants
Arm/Group | GVAX | Placebo
Number analyzed (Participants) | 30 | 27
Percentage of participants
  Grade 2-4 aGVHD @1yr | 34 | 12
  Grade 3-4 aGVHD @1yr | 16 | 0
  Chronic GVHD @3yrs | 47 | 59
  Mod-severe cGVHD @3yrs | 23 | 33

4. Secondary Outcome: Percentage of Participants With Relapse and/or Non-Relapse Mortality
Description: Percentage of participants with relapse and/or non-relapse mortality at 18 months from registration.
Time Frame: 18 Months
Measure: Number; unit: Percentage of participants
Arm/Group | GVAX | Placebo
Number analyzed (Participants) | 30 | 27
Percentage of participants
  Non-relapse Mortality | 17 | 7.7
  Relapse | 30 | 37

5. Secondary Outcome: 18-Month Overall Survival
Description: Assessment of overall survival at 18 months. Participants alive at last contact are censored at last contact.
Time Frame: 18 Month
Measure: Number; unit: Percentage of participants
Arm/Group | GVAX | Placebo
Number analyzed (Participants) | 30 | 27
Percentage of participants | 63 | 59

ADVERSE EVENTS:
Time Frame: 18 Months
Description: Patients were monitored for local and systemic adverse reactions with weekly to twice weekly examinations and laboratory studies during the study period. Acute graft-versus host disease (GVHD) was graded according to Keystone criteria.19 Non-GVHD adverse events were reported according to the National Cancer Institute Common Toxicity Criteria v.4 guidelines.
Arm/Group | GVAX | Placebo
All-Cause Mortality (participants affected / at risk) | 14/30 | 13/27
Serious Adverse Events (participants affected / at risk) | 1/30 | 2/27
Other Adverse Events (participants affected / at risk) | 10/30 | 4/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GVAX (N=30) | Placebo (N=27)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GVAX (N=30) | Placebo (N=27)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 6 | 0
Fatigue (General disorders) | 1 | 1
Skin Induration (Skin and subcutaneous tissue disorders) | 5 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/95/NCT01773395/Prot_SAP_000.pdf